CLINICAL TRIAL: NCT05636761
Title: Comparation of Heart Rate Variability Recording With Elite HRV Application and Polar V800 for the Analysis in Healthy Adults
Brief Title: Heart Rate Variability Recording With Elite HRV Application and Polar V800
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Talita Dias da Silva, Principal Investigator, University of Sao Paulo
Other Study IDs: 29108019.8.0000.5505
Record Dates: First submitted 2022-11-04; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Reliability and Validity
Keywords: Cardiovascular Risk Factors; Heart rate; Mobile Applications; Autonomic Nervous System

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group EliteHRV: the group (Elite) that started the assessment with the EliteHRV mobile application
  Interventions: Diagnostic Test: Heart rate variability
- group Polar: the (Polar) group that started the evaluation with the Polar V800 watch
  Interventions: Diagnostic Test: Heart rate variability

INTERVENTIONS:
Diagnostic Test: Heart rate variability — Collection and Analysis of Heart Rate Variability

SUMMARY:
The Elite HRV is a reliable HRV analysis tool and could be a valid option to replace the Polar V800. The objective of study is Comparing the HRV index recorded with the mobile app Elite HRV and with the multisport watch Polar V800. Individuals will submit to two RR interval recordings with a Polar H7 strap that sent the data either to the Polar V800 heart rate monitor or to the Elite HRV app. The volunteers will supine position and breathing spontaneously, and the RR intervals will collect during 25 minutes. Subsequently, without warning the subject, the strap will connect to a nother device, and the second 25minute evaluation was made. The order in which the devices will use is randomized and the HRV indexes will generated via Kubios HRV.

DETAILED DESCRIPTION:
Sample Characterization Before starting the evaluation, an anamnesis will apply, in order to know the individual characteristics of each candidate and verify if he eligible. In addition, anthropometric variables such as weight, height and Body Mass Index will perform to characterize the individuals.

Heart Rate Variability (HRV) Heart rate will recorded beat by beat using a heart rate meter (Polar H10, Polar Electro, Kempele, Finland) at a sampling rate of 5 kHz to assess cardiac autonomic modulation.

With the chest strap and the receiving and recording device (Elite HRV and Polar V800), the subjects will be positioned in the supine position and remained at rest with spontaneous breathing for 25 min. The laboratory temperature was controlled at 20°C, and data classification was performed in the morning or afternoon, always with a minimum fasting of 2 hours. Participants ask to avoid consuming coffee, chocolate or alcohol and taking medication the night before. Then, without notifying the subject, the strap will be connect to the other receiving device and a new 25-minute collection will perform.

For analysis of HRV data, the last 20 minutes of each collection will select. In the future, the first 1000 beat intervals were chosen and only series with more than 95% of sinus beats were included in the study, totaling 1000 consecutive RR intervals.

HRV analysis was performed using linear methods, analyzed in the time and frequency domains, according to the guidelines of the Task Force of the European Society of Cardiology and the North American Society of Stimulation and Electrophysiology.

STATISTICAL ANALYSIS To determine the difference between the device data, the one-sample t-test will be use. Pearson's correlation coefficient was chosen to evaluate the correlation and it was considered null, weak, moderate, strong, very strong or perfect, when, respectively, r=0; r=0 to 0.3; r=0.3 to 0.6; r=0.6 to 0.9; r=0.9 to 1; r=1.

Bland Altman Plots with limits of agreement of 95% were constructed for all indices in order to assess agreement and bias between the different forms of HRV capture. In addition, to analyze the presence of proportion bias, linear regression was used and in case of non-significance, the hypothesis of proportion bias was discarded.

We also used Multiple Analysis of Variance (MANOVA) for comparison between Groups (started with Elite HRV versus started with Polar) with Repeated Measures for comparison within Devices (Elite HRV versus Polar). ANOVA one-way with repeated measures for comparisons of Devices (without order comparison) was done to determine p value and effect size. Values of p <0.05 were considered significant. The statistical package used was the Statistical Package for Social Sciences (SPSS; IBM, Chicago, Illinois, USA), version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years of age
* Apparently healthy

Exclusion Criteria:

* Diagnoses of previously installed heart disease
* Continuous medication use that can alter HRV
* Use of any substance that could influence the autonomic nervous system, such as caffeinated drinks and foods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To determine the sample size, a sample size calculation was performed, assuming the following parameters: alpha of 5%, beta of 20% (power = 80%) and difference between groups of 10% regarding the scores on the scale. With these data, 30 subjects were calculated in each study arm.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
similarity of indices of heart rate variability between two devices | 1 day
  assessment of heart rate variability indices from both devices

CONTACTS AND LOCATIONS:
Overall Officials: Talita D da Silva, Principal Investigator — Researcher
Locations (1):
- Paulist School of Medicine, São Paulo, São Paulo, Brazil